CLINICAL TRIAL: NCT00617877
Title: Pharmacogenetic of the Antihypertensive Response to the Angiotensin II Blockers in Monotherapy or Associated to Hydrochlorothiazide
Brief Title: Antihypertensive Response to Losartan and Genetic Polymorphisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Executive Vice President, Clinical and Quantitative Sciences, Merck & Co., Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007_035; MK0954-334
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2009-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Losartan

ARMS (1):
- 1 (Experimental): Losartan 50 mg/day for 4 weeks, then doubled to losartan 100 mg/day in case of BP more than 140/90 mm Hg. HCTZ 25 mg will be added at week 8 if BP is more than 140/90 mm Hg. This last regimen will be continued until the end of the study (visit 9-week 48).
  Interventions: Drug: losartan potassium; Drug: Comparator: Hydrochlorothiazide

INTERVENTIONS:
Drug: losartan potassium — Losartan 50 mg/day for 4 weeks, then doubled to losartan 100 mg/day (in case of BP more than 140/90 mm Hg.) Continued until the end of the study (visit 9-week 48).
Drug: Comparator: Hydrochlorothiazide — Hydrochlorothiazide 25 mg will be added at week 8 if BP is more than 140/90 mm Hg. This last regimen will be continued until the end of the study (visit 9-week 48).

SUMMARY:
The purpose of this study is to evaluate the antihypertensive response of treatment with losartan with reference to genetic polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

* Both gender less than 60 years old, with mild-moderate hypertension (SBP greater than and DBP equal or greater than 90 mmhg, BP < 180/110)
* Never treated for hypertension or who have taken antihypertensive agents sporadically (not more than 15 days total therapy) but not in the 30 days prior to the first visit
* Patient in therapeutic wash out for 6 months
* Patient is asymptomatic, absence of significant concomitant diseases, except for non-familial hypercholesterolemia, absence of systemic diseases
* Women with menopause not treated with hormone replacement therapy or women of reproductive age who do not make use of estro-progestagen agents but who use another safe contraceptive method
* BMI < 30 for men and < 28 for women

Exclusion Criteria:

* Secondary or malignant hypertension, Na <130 mmol/l, K >5,5 mmol/l, or < 3,0 mmol/l
* Cardiac disease such as ischemic, HF, arrhythmia, cardiac surgery
* Pregnant, breast feeding
* History of nephropathy, metabolic disease, liver disease
* Alcohol or drug abuse
* History of angioedema
* Has a known hypersensibility to study drug(s)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 800 (Actual)
Dates: Start 2005-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Blood pressure reduction with reference to genetic polymorphisms. | Over 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC